CLINICAL TRIAL: NCT06724484
Title: Post-operative Anxiety and Depression Among Older Adults Who Undergo Surgery for Fragility Fractures
Acronym: FFAD
Status: Not yet recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 94213
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Fractures in the Elderly
Keywords: Fragility fracture; Anxiety; Depression; Surgery
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fragility fracture receiving surgery: In this group, patients who sustain a fragility fracture and receive surgical intervention will be recruited.
  Interventions: Procedure: Surgical management of fracture
- Control: In this group, patients who sustain fragility fracture and receive conservative (non-surgical) management will be recruited.
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Surgical management of fracture — Surgical management of fracture
  Groups: Fragility fracture receiving surgery
Other: No intervention — No intervention
  Groups: Control

SUMMARY:
Patients who present with falls and fractures can experience increased symptoms of depression and anxiety due to the trauma of falling, hospitalisation and surgery. Additionally after surgery, patients may be limited in their mobility, resulting in a loss in their independence which can lead to further feelings of frustration and helplessness. In this study we want to know how common this problem is among older people who are admitted to hospital with broken bones and subsequently receiving surgery.

We will use a questionnaire called the Hospital Anxiety and Depression Scale (HADS) to explore this. We will recruit 60 patients for this study, 30 participants who received operative management and a further 30 participants who did not receive surgery for comparison. Patients who are not able to consent to the study or those who are not able to complete the questionnaire will not be recruited. We will collect routine data from the patients to provide a description of the patients that we are studying. Patients will complete the HADS questionnaire once during their hospital stay and then in 1 month's time. We will contact patients through telephone for the 1 month follow up.

This study will enable us to determine how common are the symptoms of anxiety and depression among this group of patients. This will help raise awareness of the problem which may prompt further intervention and management plan to address this important issue.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and above
* Received operative or non-operative management of fragility fracture
* Able to provide written consent

Exclusion Criteria:

* Patients receiving end of life care
* Patients with known diagnosis of severe dementia and/ or lack capacity to consent
* Non-fragility fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults who are admitted to a tertiary hospital/ major trauma centre with a fragility fracture.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | This will be measured at baseline and at 1 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lim, BM, MRCP (UK), PhD, Principal Investigator — University of Southampton
Locations (1):
- Academic Geriatric Medicine, University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on the university's online repository.
Supporting Information: Study Protocol, ICF
Time Frame: Start date: September 2024 End date: August 2033
Access Criteria: Anyone who is interested in the study may be able to access the data by contacting the study PI.

REFERENCES:
- [Background] Frenkel WJ, Jongerius EJ, Mandjes-van Uitert MJ, van Munster BC, de Rooij SE. Validation of the Charlson Comorbidity Index in acutely hospitalized elderly adults: a prospective cohort study. J Am Geriatr Soc. 2014 Feb;62(2):342-6. doi: 10.1111/jgs.12635. Epub 2014 Jan 21. PMID 24521366